CLINICAL TRIAL: NCT06974838
Title: Explore the Therapeutic Effect of Theta Burst Stimulation on Emotion Regulation in Autism With Minimally Verbal Ability or Intellectual Disability
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202302085A0
Record Dates: First submitted 2025-05-14; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder; Minimally Verbal Ability; Intellectual Disability
MeSH Terms: conditions — Autism Spectrum Disorder; Intellectual Disability

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Participants received the real intervention of TBS (iTBS 1200) over the left dorsolateral prefrontal cortex for 4 weeks (5 days/week).
  *iTBS = intermittent theta burst stimulation
  Interventions: Device: intermittent theta burst stimulation
- Sham (Sham Comparator): Participants received the sham intervention of TBS (with sham coil) over the left dorsolateral prefrontal cortex for 4 weeks (5 days/week).
  Interventions: Device: intermittent theta burst stimulation

INTERVENTIONS:
Device: intermittent theta burst stimulation — stimulatory protocol

SUMMARY:
The investigator would like to investigate the impact of theta-burst stimulation over left DLPFC in autism with minimally verbal ability or intellectual disability

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism spectrum disorder, confirmed by DSM-5.
* Individuals with minimal verbal ability or intellectual disability (FSIQ < 70).

Exclusion Criteria:

* Current or past severe neurological disorders, such as epilepsy, or significant visual or hearing impairments.
* Current or past severe systemic diseases, such as cardiovascular disease, diabetes, or multiple sclerosis.
* History of severe brain injury.
* Presence of implanted metal devices, such as a pacemaker or medication pump.
* Current or past severe psychiatric disorders, such as schizophrenia, bipolar disorder, or major depressive disorder.
* Pregnancy.
* Significant brain abnormalities, such as intracranial space-occupying lesions.
* Family history of epilepsy.
* History of febrile seizures.
* Concurrent use of medications that increase the risk of seizures.
* Sleep disorders during rTMS procedures.
* Skin lesions or trauma at the stimulation site.
* Deemed ineligible by the principal investigator (PI).
* Participation in another clinical trial within the past month.
* Suicidal ideation or suicide attempts within the past year.

Ages: 8 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-26 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Total Scores of Aberrant Behavior Checklist | Baseline, Week 4, Week 8 and Week 12
  Aberrant Behavior Checklist is a parents' report questionnaire for aberrant behavior. The lower scores stand for less aberrant behavior.
Total Scores of Emotional Dysregulation Inventory | Baseline, Week 4, Week 8 and Week 12
  Emotional Dysregulation Inventory is a parents' report questionnaire for emotional dysregulation. The lower scores stand for better emotional regulation.
Total Scores of Child Behavior Checklist | Baseline, Week 4, Week 8 and Week 12
  Child Behavior Checklist is a parents' report questionnaire for behavioral and emotional problems. The lower scores stand for better behavioral and emotional regulation.

SECONDARY OUTCOMES:
Total Scores of Social Responsiveness Scale | Baseline, Week 4, Week 8 and Week 12
  Social Responsiveness Scale can measure the autism clinical severity. The lower scores stand for better social responsiveness.
Total Scores of Repetitive Behavior Scale-Revised | Baseline, Week 4, Week 8 and Week 12
  Repetitive Behavior Scale-Revised is a questionnaire that focuses on repetitive behavior. The lower scores stand for lower repetitive behavior.
Total Scores of Adaptive Behavior Assessment System | Baseline, Week 4, Week 8 and Week 12
  Adaptive Behavior Assessment System is a parents' report questionnaire for adaptive behavior. The higher scores stand for better adaptive behavior.
Total Scores of Anxiety, Depression, and Mood Scale | Baseline, Week 4, Week 8 and Week 12
  Anxiety, Depression, and Mood Scale is a parents' report questionnaire for mental disorders (manic/ hyperactive behavior, depressed mood, social avoidance, general anxiety, obsessive/compulsive behavior) . The higher scores stand for higher mental problem.
Accuracy of Frith-Happe Animation | Baseline, Week 4, Week 8 and Week 12
  A quick and objective test of Theory of Mind. 8 questions in total, the more correct questions stand for better Social Cognition.
Accuracy of Eyes Task | Baseline, Week 4, Week 8 and Week 12
  An advanced test for Theory of Mind. 43 questions in total, the more correct questions stand for better social skills.
Accuracy of Wisconsin Card Sorting Test | Baseline, Week 4, Week 8 and Week 12
  An advanced test for cognitive flexibility. 128 questions in total, the more correct questions stand for better cognitive flexibility.
Accuracy of Raven's Progressive Matrices | Baseline, Week 4, Week 8 and Week 12
  An advanced test for for executive function. 60 questions in total, the more correct questions stand for better executive function.
Total Scores of Behavior Rating Inventory of Executive Function | Baseline, Week 4, Week 8 and Week 12
  Behavior Rating Inventory of Executive Function is a parents' report questionnaire for executive function. The lower scores stand for better executive function.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan